CLINICAL TRIAL: NCT01995422
Title: Effects of Physical Activity Program on the Emotional and Cognitive Dynamics in Major Depressive Disorder Patients
Brief Title: Effect of Physical Activity on Depressive Symptoms With a 5 Month Follow-up
Acronym: 2DPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratory Motricité, Interactions, Performance (Other)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-A00934-37
Record Dates: First submitted 2013-11-12; First posted 2013-11-26 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Follow-up study; Ecological momentary assessment; Physical activity; Depression; Self-esteem; Anxiety; Rumination; Quality of life
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity; Depression; Anxiety Disorders; Rumination Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical activity program (Experimental): A 5-month follow-up including a 3-month period of supervised physical activity
  Interventions: Other: Physical activity program

INTERVENTIONS:
Other: Physical activity program — One hour sessions of active walking occurring three times a week during three months

SUMMARY:
The main objective of this study is to evaluate the effect of a 12 weeks adapted physical activity program (active walking) on depression by analyzing the dynamics of emotional and cognitive functioning. The secondary objectives are to test the effects of a physical activity on functional performance and to highlight psychological mechanisms.

DETAILED DESCRIPTION:
Primary outcomes:

Self evaluations concerning global self-esteem, a perception of competence and satisfaction in the physical self and four sub-domains that are perceived physical endurance, perceived competence in sports, perceived physical force and perceived physical appearance, are performed.

Assessment of depressive symptomatology is also realised including momentary levels of depression, anxiety, rumination, efficacy of coping strategies and quality of life.

Secondary outcomes:

Assessment of postural control

ELIGIBILITY:
Inclusion Criteria:

* Speaking French
* Aged between 18 and 65 years
* Diagnosed with current major depressive disorder
* BDI II score ≥ 12
* IPAQ score <600

Exclusion Criteria:

* Alcohol or substance(s) dependence(s)
* Psychotic disorders
* Anti-social personality
* Pregnant or nursing women
* Physical inability to perform active walking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effect of physical activity on depression | Five months
  Evaluate the evolution of depressive symptoms in middle to severe depressive patients during a physical activity program

SECONDARY OUTCOMES:
Distraction, self-efficacy and social support scores on 7-point Likert scales and balance on force platform | Five months
  Exploration of underlying mechanisms associated with an expected decrease of depressive symptoms after a physical activity program concerning functional and psychological processes

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bourbousson, PhD, Study Director — Laboratory MIP
Locations (1):
- University of Nantes, Nantes, Pays de la Loire Region, France

REFERENCES:
- [Derived] Deschamps T, Thomas-Ollivier V, Sauvaget A, Bulteau S, Fortes-Bourbousson M, Vachon H. Balance characteristics in patients with major depression after a two-month walking exercise program: A pilot study. Gait Posture. 2015 Oct;42(4):590-3. doi: 10.1016/j.gaitpost.2015.07.057. Epub 2015 Jul 31. PMID 26260007